CLINICAL TRIAL: NCT00373048
Title: Mefloquine Malaria Prophylaxis in HIV-1 Infected Individuals and Its Influence on the Evolution Towards AIDS: a Randomized Placebo-controlled Trial
Brief Title: Mefloquine Prophylaxis in HIV-1 Individuals: a Randomized Placebo-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Professor Umberto D'Alessandro, Institute of Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Mefloquine HIV zambia
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: HIV Infections
Keywords: HIV-1 malaria Clinical Trial
MeSH Terms: conditions — HIV Infections | interventions — Mefloquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo, tablet (Placebo Comparator)
  Interventions: Drug: placebo
- mefloquine, tablet (Experimental)
  Interventions: Drug: mefloquine

INTERVENTIONS:
Drug: mefloquine — tablet, once weekly
  Arms: mefloquine, tablet
Drug: placebo — tablet, once weekly
  Arms: Placebo, tablet

SUMMARY:
This is a randomized placebo controlled trial. Malaria chemoprophylaxis with mefloquine in asymptomatic HIV-infected adults living in a malaria endemic region of Luanshya, Zambia will be compared to a placebo control group and followed up for 18 months.

DETAILED DESCRIPTION:
In Zambia prompt treatment of malaria cases is the mainstay of malaria control; antimalarial chemoprophylaxis is not currently recommended for general use so that the use of placebo as a comparator in this study is justified. We will analyse safety and efficacy of mefloquine, malaria and AIDS related parameters at predefined time points, and verify if this intervention could produce a slower decrease in CD4 counts compared to passive case management of malaria.

This is a randomized placebo controlled trial. Malaria chemoprophylaxis with mefloquine in asymptomatic HIV-infected adults living in a malaria endemic region of Luanshya, Zambia will be compared to a placebo control group and followed up for 18 months.

Specific designed studies taking into account possible confounding parameters (and interactions) are needed to measure the impact of malaria control in an HIV endemic environment. In particular, the question should be answered if malaria control has an impact on the disease progression of HIV. The possible impact of these interventions on morbidity and mortality taking into account these parameters might have a major public health impact. This might be on the use of antiretroviral drugs, the incidence of clinical (eventually severe) malaria and spread of antimalarial resistance through immune compromised HIV patients (with and without antimalarial treatment).

Studies of alternative strategies that contribute (next to antiretrovirals) to the control and prevention of HIV pandemic are equally important and urgently needed. The need to design these strategies is critical given the high incidence of malaria and HIV in countries in Sub Saharan Africa such as Zambia and its serious impact on survival and the socio-economic situation. Moreover, a cost-benefit analysis might show that some alternative strategies have a major impact on the field with less technical, financial and social constraints than the strategies recommended so far.

All HIVP patients will be treated for opportunistic infections (OI) and receive antiretroviral drugs following the National guidelines on Management and Care of Patients with HIV/AIDS (also if this occurs after the study period). At the time they need cotrimoxazole prevention or/and receive antiretrovirals they would have reached a study endpoint and will be excluded from the trial though the follow up will continue.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents of the Luanshya district
* Males and non pregnant adults between 18 and 50 years old.
* Having a CD4 cell count of least 350 perµL at enrolment
* HIV sero-status determined at the VCT of the health center.
* No obvious underlying disease at time of enrolment
* Signed informed consent

Exclusion Criteria:

* HIV stage III or IV following the WHO classification (see attached documents regarding policy in Zambia)
* Evidence of underlying chronic diseases (cardiac, renal, hepatic, malnutrition, TB).
* Intent to move out of the study catchment area during the study period
* History of allergy to MQ (or related drugs) or sulfa drugs
* Chorionic gonadotrophic hormone in urine or obvious pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Rate of decline of CD4 counts between different time points | months 0, 6, 12 and 18
Proportion of patients entering the AIDS stage (WHO stage 3,4) | during 18 months

SECONDARY OUTCOMES:
Mean difference in log plasma viral load at different time points, | during 18 months
Rate of decline of humoral immunity between different time points. | during 18 months
Proportion of patients with parasitaemia at the end of the intervention. | during 18 months
All cause disease incidence and prevalence (including malaria, TB) | during 18 months
Proportion of patients with Adverse event during monitoring | during 18 months
Prevalence of anaemia at different time points | during 18 months
Incidence of severe anaemia | during 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'Alessandro, MD,MSc, PHD, Study Director — Institute of Tropical Medicine Antwerp
Locations (1):
- Tropical Disease Research Center, Ndola, Cupperbelt, Zambia